CLINICAL TRIAL: NCT02851017
Title: Exergaming (XBOX Kinect™) Versus Traditional Gym-based Exercise for Postural Control, Flow and Technology Acceptance in Healthy Adults: a Randomised Controlled Trial
Brief Title: Exergaming Versus Gym-based Exercise for Postural Control, Flow and Technology Acceptance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Teesside University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HLS-GB-17-7-16
Record Dates: First submitted 2016-07-27; First posted 2016-08-01 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Young Adults
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exergaming group (XBOX Kinect (Experimental): Kinect™ exercise group performed sessions on three non-consecutive days per week for 4 weeks (12 sessions in total).
  Interventions: Other: Exercise
- Traditional gym based exercise group (Experimental): Traditional gym based (TGB) exercise group performed sessions on three non-consecutive days per week for 4 weeks (12 sessions in total). Those in the TGB group performed exercises that were matched for sequence, intensity, duration and mode of exercise by adopting open and closed kinetic chain movements, in the same range and loading as required in the Kinect™ group.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — This study is designed to examine and comparing there intervention program on postural control, flow and technology acceptance in young healthy adults.

SUMMARY:
Balance training is an important component of physical fitness, however due to the mundane and often repetitive nature of balance training alone this is often forgotten about and as a result people may be more susceptible to postural control instabilities. A potential solution to the mundane aspect of balance training is the use of exergaming (interactive exercise and gaming combined) through the use of commercial gaming systems such as the Nintendo Wii, Dance Dance Revolution (DDR) and more recently the XBOX Kinect. The aim of the investigation was to assess the XBOX Kinect versus traditional balance training on postural control, flow and technology acceptance.

DETAILED DESCRIPTION:
Exergaming - exercise with the use of an interactive computer-generated environment - is increasingly used in physical rehabilitation. Benefits have been reported in a range of clinical populations (people with neurological problems children with cerebral palsy and learning difficulties, Parkinson' disease, multiple sclerosis and older people. Balance training is an important focus of such rehabilitation. Previous literature regarding the effects of exergaming as a method of balance-training has mainly been conducted using the Nintendo Wii™ and the Wii™ fit where people must stand on a balance board to play the games. Although literature has shown that traditional balance training alone is effective in improving balance in a range of populations, studies comparing exergaming with "traditional" balance exercises (SEBT, trampolines and wobble boards) have shown mixed results from both exergaming and traditional balance training groups improving in postural control outcomes to greater improvement in the exergaming group over traditional balance exercise. A potential reason for the differentiation if results could be due to different movements required in the "traditional" balance exercises rather than there being something inherently different about exercising in a virtual environment. There is also a dearth of randomized controlled trials (RCT) in this area so the evidence base is limited. Furthermore, few have studied the important psychological aspect of exergaming, in particular acceptance and flow experience. The aim of this study was to assess the effects of exergaming using the XBOX Kinect™ system, versus, traditional gym-based exercise, with no virtual stimuli (TGB) on: (1) postural control, (2) technology acceptance (3) flow experience and (4) exercise intensity in young healthy adults. Matching of intensity of exercise, in the two groups, was assessed objectively, by Heart Rate and subjectively by Borg RPE during all exercise sessions. To our knowledge this is the first paper to compare the effects of exergaming against matched traditional exercises where the movement patterns, intensity and physiological demand was matched and assessed across groups.

ELIGIBILITY:
Inclusion Criteria:

* Male or female,
* Aged 18-50 years,
* Physically active (three or more moderate-vigorous physical activity sessions per week), free from injury (no musculoskeletal injuries or neurological conditions)
* Able to take part in four weeks of exercise.

Exclusion Criteria:

* Unable to give informed consent and/or to comprehend and write English,
* Current (or history of) any medical condition or injury which would contraindicate participation,
* Allergy to alcohol wipes and/or adhesive tape
* Previous experience of using the XBOX Kinect™.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Postural control | Change from baseline (week 1) to post intervention (week 4)
  Postural sway was measured using a portable Kistler™ force platform (Model 9286AA, W 40 x L 60 x H 3.5cm). Participants were instructed to stand as still as possible with their arms by their side and eyes open, on their dominant leg (preferred kicking) for five periods of 30 seconds. Between trials, participants stepped off the force plate to allow calibration of the equipment which gave a 30 seconds rest.
Flow State Scale | Change from baseline (week 1) to post intervention (week 4)
  The questionnaire consist of a 36-item questionnaire with nine subscales and response options on a Likert scale from 1 (strongly disagree) to 5 (strongly agree). Dimensions of flow include challenge-skill balance (CB; skills match the task and will be successful); clear goals (CG; experience of having a pre-set goal which on is aiming to achieve); unambiguous feedback (UF; feedback on performance); concentration of task (CT; focused on task); paradox of control (PC; performs task with ease); action-awareness-merging (AM; automatic response to task); transformation of time (TT; time speeds up or slows down during activity); loss of self-consciousness (LS; immersed in task) and autotelic experience (AE; activity intrinsically rewarding).
Unified Theory of Acceptance and Use of Technology (UTAUT) | Change from baseline (week 1) to post intervention (week 4)
  Technology acceptance was measured using UTAUT which comprised a 7-point Likert scale, with response options on a Likert scale from 1 (strongly disagree) to 7 (strongly agree). The questionnaire has six main domains, performance expectancy (PE; system will help performance), Effort Expectancy (EE; ease of using system), Social Influence (SI; degree in which others believe they should use system), Facilitating Conditions (FC; support in using the system), Self-efficacy (SE; confidence in using the system) and Behavioural Intention (BI; intention to use the system again).

SECONDARY OUTCOMES:
Heart Rate | Change from baseline (week 1) to post intervention (week 4)
  Heart rate (HR) was recorded using a Polar™ Heart Rate Monitor™ (FS2C), recording watch and T31 coded chest strap (Polar Electro, Oy, Finland). Mean HR was collected at the end of every exercise session and calculated as a percentage of predicted HR max (220 - age).
BORG subjective exertion scale | Change from baseline (week 1) to post intervention (week 4)
  For a subjective measure of physiological cost the BORG Rate of Perceived Exertion (RPE) scale was used. Mean RPE data were recorded in each exercise session. RPE was defined as how hard participants felt their body was working in general based on the physical sensations they may experience during the activity, including increases in HR, respiration, breathing rate, sweating, and muscle fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Gill Barry, PhD, Principal Investigator — Northumbria University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Esculier JF, Vaudrin J, Beriault P, Gagnon K, Tremblay LE. Home-based balance training programme using Wii Fit with balance board for Parkinsons's disease: a pilot study. J Rehabil Med. 2012 Feb;44(2):144-50. doi: 10.2340/16501977-0922. PMID 22266676
- [Background] dos Santos Mendes FA, Pompeu JE, Modenesi Lobo A, Guedes da Silva K, Oliveira Tde P, Peterson Zomignani A, Pimentel Piemonte ME. Motor learning, retention and transfer after virtual-reality-based training in Parkinson's disease--effect of motor and cognitive demands of games: a longitudinal, controlled clinical study. Physiotherapy. 2012 Sep;98(3):217-23. doi: 10.1016/j.physio.2012.06.001. Epub 2012 Jul 9. PMID 22898578
- [Background] Saposnik G, Teasell R, Mamdani M, Hall J, McIlroy W, Cheung D, Thorpe KE, Cohen LG, Bayley M; Stroke Outcome Research Canada (SORCan) Working Group. Effectiveness of virtual reality using Wii gaming technology in stroke rehabilitation: a pilot randomized clinical trial and proof of principle. Stroke. 2010 Jul;41(7):1477-84. doi: 10.1161/STROKEAHA.110.584979. Epub 2010 May 27. PMID 20508185
- [Background] Bryanton C, Bosse J, Brien M, McLean J, McCormick A, Sveistrup H. Feasibility, motivation, and selective motor control: virtual reality compared to conventional home exercise in children with cerebral palsy. Cyberpsychol Behav. 2006 Apr;9(2):123-8. doi: 10.1089/cpb.2006.9.123. PMID 16640463
- [Background] Weiss PL, Bialik P, Kizony R. Virtual reality provides leisure time opportunities for young adults with physical and intellectual disabilities. Cyberpsychol Behav. 2003 Jun;6(3):335-42. doi: 10.1089/109493103322011650. PMID 12855092
- [Background] Pompeu JE, Mendes FA, Silva KG, Lobo AM, Oliveira Tde P, Zomignani AP, Piemonte ME. Effect of Nintendo Wii-based motor and cognitive training on activities of daily living in patients with Parkinson's disease: a randomised clinical trial. Physiotherapy. 2012 Sep;98(3):196-204. doi: 10.1016/j.physio.2012.06.004. Epub 2012 Jul 25. PMID 22898575
- [Background] Robinson J, Dixon J, Macsween A, van Schaik P, Martin D. The effects of exergaming on balance, gait, technology acceptance and flow experience in people with multiple sclerosis: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2015 Apr 17;7:8. doi: 10.1186/s13102-015-0001-1. eCollection 2015. PMID 25969739
- [Background] Van Schaik P, Blake J, Pernet F, Spears I, Fencott C. Virtual augmented exercise gaming for older adults. Cyberpsychol Behav. 2008 Feb;11(1):103-6. doi: 10.1089/cpb.2007.9925. PMID 18275322
- [Background] Venkatesh V, Morris M, Davis G, Davis F. User acceptance of information technology: toward a unified view. Management Information Systems Quarterly. 27:425-78, 2003.
- [Background] Jackson SA, Marsh H. Development and validation of a scale to measure optimal experience: The Flow State Scale. J Sport and Exercise Psychology. 18:17-35, 1996.
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Derived] Barry G, van Schaik P, MacSween A, Dixon J, Martin D. Exergaming (XBOX Kinect) versus traditional gym-based exercise for postural control, flow and technology acceptance in healthy adults: a randomised controlled trial. BMC Sports Sci Med Rehabil. 2016 Aug 23;8(1):25. doi: 10.1186/s13102-016-0050-0. eCollection 2016. PMID 27555917